CLINICAL TRIAL: NCT00014092
Title: Treatment of Patients With Metastatic Malignant Melanoma With Chemobiotherapy With Temozolomide, GM-CSF, IL2, and Interferon Alfa-2b Phase II Trial
Brief Title: Chemotherapy Followed by Biological Therapy in Treating Patients With Stage IV Melanoma That Cannot be Treated With Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saint Francis Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067958; SFMH-BB-IND-5301; NCI-V00-1591
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2004-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interferon-alpha; sargramostim; Temozolomide

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as interleukin-2 and interferon alfa stimulate a person's white blood cells to kill cancer cells or may interfere with the growth of cancer cells. Combining chemotherapy with biological therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of temozolomide followed by sargramostim, interleukin-2, and interferon alfa in treating patients who have stage IV melanoma that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, time to progression, and survival of patients with unresectable stage IV melanoma treated with temozolomide followed by sargramostim (GM-CSF), interleukin-2, and interferon alfa.
* Determine the safety and tolerability of this regimen in this patient population.
* Determine the changes in quality of life over time in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide on days 1-5, and sargramostim (GM-CSF), interleukin-2, and interferon alfa subcutaneously on days 6-17. Treatment repeats every 28 days for 4-8 courses in the absence of disease progression or unacceptable toxicity. Patients with at least stable or responsive disease after 8 courses of therapy may receive additional therapy at investigators discretion.

Quality of life is assessed at baseline, every 8 weeks during study, and then at 1 month after study.

Patients are followed at 1 month, every 3 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable stage IV melanoma
* Measurable metastatic disease
* No uncontrolled brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* BUN no greater than 1.5 times ULN
* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No significant cardiovascular disease

Other:

* No non-malignant systemic disease
* No acute infection requiring IV antibiotics
* No alcohol or substance abuse
* No other condition, disease, or history of other illness that would preclude study participation
* No hypersensitivity, allergic reactions, or intolerance to study drugs
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No prior interleukin-2
* No other concurrent immunotherapy
* No concurrent investigational vaccines or immunomodulatory agents
* No other concurrent growth factors

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No prior temozolomide
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent steroids (including corticosteroids)

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior major surgery

Other:

* At least 30 days since prior immune-based therapy
* No concurrent participation in other clinical trials with investigational drugs
* No other concurrent anticancer drugs
* No concurrent immunosuppressive therapy
* No concurrent levamisole or cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Spitler, MD, Study Chair — Northern California Melanoma Center at St. Francis Memorial Hospital
Locations (3):
- United States (3):
  - Saint Francis Memorial Hospital, San Francisco, California
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado

REFERENCES:
- [Result] Weber RW, O'Day S, Rose M, Deck R, Ames P, Good J, Meyer J, Allen R, Trautvetter S, Timmerman M, Cruickshank S, Cook M, Gonzalez R, Spitler LE. Low-dose outpatient chemobiotherapy with temozolomide, granulocyte-macrophage colony stimulating factor, interferon-alpha2b, and recombinant interleukin-2 for the treatment of metastatic melanoma. J Clin Oncol. 2005 Dec 10;23(35):8992-9000. doi: 10.1200/JCO.2005.02.5791. Epub 2005 Oct 31. PMID 16260693